CLINICAL TRIAL: NCT02538809
Title: Quantitative Evaluation of a Novel mRNA-based Urine Test for Bladder Cancer in Spinal Cord Individuals With Symptoms or Clinical Findings Suspicious for Bladder Cancer
Brief Title: Novel mRNA-based Urine Test for Bladder Cancer in Spinal Cord Injury Individuals
Status: Terminated | Type: Observational
Why Stopped: insufficient recruitment
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Sponsor
Other Study IDs: 2014-21-v2
Record Dates: First submitted 2015-08-27; First posted 2015-09-02 (Estimated); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Bladder Cancer; Spinal Cord Injury
MeSH Terms: conditions — Urinary Bladder Neoplasms; Spinal Cord Injuries | interventions — Urination

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: measurement of tumor mRNA concentration in urine — bed-side test of tumor mRNA concentration in urine

SUMMARY:
Bladder cancer is a well-recognized complication in spinal cord injury (SCI) individuals. The observed incidence rates in SCI individuals are considerably higher compared to the general population. Bladder cancer in SCI individuals tends to present at an earlier age compared to the general population. Furthermore, bladder cancer in SCI individuals is more commonly invasive and at a more advanced stage at the time of diagnosis compared to bladder cancer in the general population. Individuals with bladder cancer commonly present with hematuria and other urinary symptoms. The gold standard for diagnosis is cystoscopy. However in SCI individuals, hematuria may get attributed to catheter irritation or trauma or an urinary tract infection. Furthermore, the bladder wall commonly presents with various changes under cystoscopic examination masking the presence of a bladder wall mass. Thus, diagnosis of bladder cancer in SCI individuals can be complicate.

There is a novel test available (GeneXpert® Bladder Cancer Detection, Cepheid International, Sunnyvale, CA, USA) for the measurement of mRNA bladder tumor markers in the urine. The diagnostic accuracy of this test has been investigated in non-SCI individuals with symptoms suspicious for bladder cancer. The test showed high sensitivity and specificity values and is thus a promising diagnostic or screening tool.. However, the diagnostic accuracy of the test has not yet been investigated in SCI individuals.

The primary objective of the proposed study is to investigate whether urine mRNA tumor marker levels in spinal cord injury individuals with symptoms and findings suspicious for bladder cancer are a discriminator between individuals suffering from bladder cancer and those not suffering from cancer.

Individuals presenting with symptoms suspicious of bladder cancer will undergo ultrasonic and cystoscopic examination of the bladder. An urine sample will be taken, and the bladder will be flushed for collecting a bladder fluid sample. In patients with bladder wall findings suspicious of cancer, a bladder wall biopsy will be taken, according to clinical standard practice. The bladder fluid and the bladder wall biopsy will be submitted for cytology and histopathology examination, respectively. Tumor mRNA levels will be measured in the urine sample.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms suspicious of bladder cancer (haematuria, ultrasonic and cystoscopy findings)
* Chronic spinal cord injury for a minimum of 3 years
* Informed Consent as documented by signature

Exclusion Criteria:

* Age < 18 years
* History of bleeding disorder
* Bladder augmentation
* Acute, symptomatic urinary tract infection
* Pregnancy
* Urolithiasis
* Previous intravesical treatment (e.g. bladder irrigation, botulinum toxin injection) < 2 weeks)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: individuals presenting with symptoms or clinical findings suspicious for bladder cancer at a tertiary urologic referral center
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
urine tumor mRNA concentration | 1 day

SECONDARY OUTCOMES:
cystoscopic findings of bladder wall | 1 day
  findings suspicious of bladder cancer present: yes / no
microscopic identification of cells in bladder fluid sample | 1 day
histopathologic examination of the bladder wall biopsy | 1 day
  diagnosis of bladder cancer: yes / no

CONTACTS AND LOCATIONS:
Overall Officials: Jens Wöllner, Principal Investigator — Schweizer Paraplegiker-Zentrum Nottwil
Locations (1):
- Swiss Paraplegic Centre, Nottwil, Canton of Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No